CLINICAL TRIAL: NCT07067684
Title: The Effect of Low Tidal Volume Ventilation on Diaphragmatic Excursion in Cardiopulmonary Bypass Surgery
Brief Title: LTV (Low Tidal Volüme) Ventilation and Diaphragmatic Motion in CABG (Coronary Artery Bypass Grafting)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Nuran Akıncı Ekinci, MD, Anesthesiologist, Department of Anesthesiology, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Diaflex
Record Dates: First submitted 2025-07-02; First posted 2025-07-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-08

CONDITIONS: Perioperative Respiratory Function; Diaphragmatic Dysfunction; Low Tidal Volume Ventilation
Keywords: Low Tidal Volume Ventilation; Diaphragmatic Excursion; Coronary Artery Bypass Grafting (CABG)

STUDY DESIGN:
Intervention Model Description: randomized, controlled, parallel-assignment trial with an assessor-blinded design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only participants and outcome assessors are masked in this study. No additional masked parties beyond those listed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Low (Experimental): Low Tidal Volume Ventilation Group (LTV)
  Interventions: Other: Low Tidal Volume Ventilation During CPB
- Group Apnea (No Intervention): Apnea Group (Control Group)

INTERVENTIONS:
Other: Low Tidal Volume Ventilation During CPB — Group Low: Patients in this group will receive low tidal volume mechanical ventilation during cardiopulmonary bypass (CPB).
  Ventilation settings will be:
  Tidal Volume: 3-4 mL/kg (ideal body weight)
  PEEP: 5-8 cmH₂O
  Respiratory Rate: adjusted to maintain normocapnia (PaCO₂ 35-45 mmHg)
  Arms: Group Low

SUMMARY:
The goal of this clinical trial is to evaluate whether low tidal volume (LTV) ventilation during cardiopulmonary bypass (CPB) surgery helps preserve diaphragmatic excursion in adult patients undergoing coronary artery bypass grafting (CABG). The study will also assess the relationship between LTV ventilation and postoperative pulmonary complications, such as atelectasis, pleural effusion, and pneumonia.

The main questions this trial aims to answer are:

Does LTV ventilation better preserve diaphragmatic motion compared to apnea during CPB?

Are postoperative pulmonary complications less frequent in patients receiving LTV?

Does LTV contribute to shorter extubation times and ICU stays?

Researchers will compare LTV ventilation with apnea (standard care) during CPB to assess its effects on diaphragmatic excursion, measured via ultrasound, and postoperative respiratory outcomes.

Participants will:

Undergo elective CABG surgery under general anesthesia

Be randomly assigned to receive either LTV ventilation or apnea during CPB

Have diaphragmatic excursion measured by ultrasound before surgery, before extubation, and 24 hours after surgery

Be monitored for postoperative pulmonary complications (atelectasis, effusion, pneumonia), extubation time, and ICU length of stay

Ultrasound will be used to measure diaphragmatic excursion (DE) in quiet and deep breathing. DE below 10 mm will be considered as diaphragmatic paralysis. Postoperative respiratory assessments will include blood gas analysis (PaO₂/FiO₂ ratio), clinical respiratory parameters, and imaging findings.

This is a prospective, single-center, assessor-blinded randomized controlled trial. Patients and outcome assessors will be blinded to group allocation. The study will be conducted at the Anesthesiology Clinic of Konya City Hospital and is expected to enroll 60 patients.

DETAILED DESCRIPTION:
oronary artery bypass grafting (CABG) surgery performed under cardiopulmonary bypass (CPB) is a complex procedure frequently associated with postoperative pulmonary complications (PPCs). During CPB, mechanical ventilation is usually paused (apnea), which leads to temporary diaphragmatic inactivity. The diaphragm, being a rhythmically contracting muscle under normal physiological conditions, may experience transient dysfunction or even paralysis due to this intraoperative inactivity. Several mechanisms, including loss of neuromechanical coupling, disrupted neuromuscular signaling, altered venous return, and impaired diaphragmatic oxygenation and metabolism, are thought to contribute to this process.

Reduced diaphragmatic motion can create a favorable condition for atelectasis, impair oxygenation, and increase the risk of infection in the postoperative period. The resulting transient diaphragmatic dysfunction is considered a potential contributor to the development of PPCs such as pneumonia, pleural effusion, and prolonged mechanical ventilation.

Recent research has focused on the protective effects of low tidal volume (LTV) ventilation in surgical and critical care settings. However, limited studies have evaluated its direct impact on diaphragmatic function during CPB, particularly in the context of CABG surgery. There is a need to investigate whether intraoperative application of LTV ventilation during CPB can help preserve diaphragmatic excursion (DE) and reduce PPCs.

ELIGIBILITY:
Inclusion Criteria:

Age over 18 years

Male or female patients

American Society of Anesthesiologists (ASA) physical status class II or III

Scheduled for elective coronary artery bypass graft (CABG) surgery with cardiopulmonary bypass (CPB)

Provided written informed consent to participate in the study -

Exclusion Criteria:

History of neuromuscular disease

History of thoracic surgery

History of pneumothorax or ascites

Chronic respiratory failure

Pulmonary hypertension or right ventricular failure

Emergency surgery

Inability to perform diaphragm ultrasonographic measurements

Refusal to participate in the study

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Diaphragmatic Excursion Measured by Ultrasound | Baseline (30 minutes before transfer to the operating room (Preoperative baseline) Postoperative ( Immediately Before Extubation) 24 Hours After Surgery (24 hours after the end of surgery)
  Diaphragmatic excursion (DE) will be measured using M-mode ultrasonography with a 2-5 MHz convex probe placed in the anterior subcostal view. Measurements will be performed during both quiet and deep breathing maneuvers. A DE value of ≤10 mm will be considered indicative of diaphragmatic paralysis. The average of three consecutive measurements will be recorded at each time point. The main comparison will assess postoperative DE values between groups receiving low tidal volume ventilation and apnea during CPB.

SECONDARY OUTCOMES:
Incidence of Postoperative Pulmonary Complications | First 3 Days After Surgery and Prior to ICU Discharge
Time to Extubation | From ICU Admission to Extubation (Up to 24 Hours Postoperatively)
  The time from ICU admission to successful extubation will be recorded in hours. Extubation will be performed based on predefined weaning criteria, including neurological status, respiratory stability, hemodynamic parameters, and oxygenation status. Patients not meeting criteria within 24 hours will be recorded accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The plan to share individual participant data has not been determined. No data will be shared at this stage due to institutional policy and ethical concerns.

REFERENCES:
- [Result] Barbariol F, Deana C, Guadagnin GM, Cammarota G, Vetrugno L, Bassi F. Ultrasound diaphragmatic excursion during non-invasive ventilation in ICU: a prospective observational study. Acta Biomed. 2021 Jul 1;92(3):e2021269. doi: 10.23750/abm.v92i3.11609. PMID 34212900